CLINICAL TRIAL: NCT02446223
Title: A Pilot Prospective Clinical Trial to Evaluate the Efficacy and Safety of Large-Scale, Field-Directed Topical Therapy of Actinic Keratosis of the Chest With Ingenol Mebutate 0.015%
Brief Title: Evaluate the Efficacy and Safety of Large-Scale Field-Directed Topical Therapy of Actinic Keratosis of the Chest w/Ingenol Mebutate 0.015%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PICATO-2013-01
Record Dates: First submitted 2015-05-12; First posted 2015-05-18 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis AKs Chest Pre-Cancer
MeSH Terms: conditions — Keratosis, Actinic

ARMS (1):
- Active (Experimental)
  Interventions: Drug: Inggenol Mebutate 0.015%

INTERVENTIONS:
Drug: Inggenol Mebutate 0.015%

SUMMARY:
Evaluate the Efficacy and Safety of Large-Scale Field-Directed Topical Therapy of Actinic Keratosis of the Chest w/Ingenol Mebutate 0.015%

DETAILED DESCRIPTION:
This will be an open-label study to evaluate the efficacy and safety of ingenol mebutate gel, 0.015% used in topical therapy of actinic keratosis on the chest. Subjects that present with 4 or more actinic keratosis in one continuous 100cm2 area of the chest and meet all inclusion/exclusion criteria will be enrolled into this study.

Treatment with the investigational product (IP) will be applied for three continuous days. The investigator will guide application of the IP in-office at Day 0 and the subject will be instructed to self-administer the IP at Days 1 and 2. Follow-up visits will be scheduled at Days 1, 3, 10, 17, 24 and 59.

Prior to treatment and at each visit, the investigator will assess the subject's treatment area for lesion counts and at follow up visits 4, 5, 6 and 7 evaluation of clearance. Pre-treatment photography will also be collected at baseline and at each follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of at least 18 years of age.
2. Subjects willing to comply with study requirements.
3. The presence of four or more clinically typical actinic keratosis within one contiguous area of the chest that is 100cm2.
4. For female subjects of childbearing potential willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use at least 30 days prior to entry into the study.

   A female is considered NOT to be of childbearing potential if she is postmenopausal for at least one (1) year, without a uterus, without both ovaries or has had a bilateral tubal ligation.

   Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants Norplant, Depo-Provera, double-barrier methods (e.g. condoms and spermicide) and abstinence.
5. Subjects willing to refrain from the use of topical products containing alpha-hydroxy acids, retinoic acid, retinol, salicylic acid, and vitamins C/D (or their derivatives) in the treatment area 7 Days prior to and during the entire study period

Exclusion Criteria:

1. Known hypersensitivity, prior allergic reaction, or prior chest treatment with ingenol mebutate gel.
2. Treatment area containing hypertrophic or hyperkeratotic lesions, cutaneous horns or lesions that had previously not responded to other standard treatments.
3. Presence of any skin condition or disease that might interfere with the diagnosis and evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis, seborrheic dermatitis).
4. Subjects receiving ablative laser treatments on their chest must have discontinued the treatment at least 6 months prior to entering the study.
5. Subjects receiving Intense Pulse Light treatments on their chest must have discontinued the treatment at least 30 days prior to entering the study.
6. Within 3 months of study entry treatments that may interfere with evaluation of the treatment area (e.g. other topical therapies for actinic keratosis of the chest, topical corticosteroids, topical retinoids, ultraviolet B phototherapy, or immunosuppressive, immunomodulating, or cytotoxic medications) or expected use of any of the above-mentioned therapies in the treatment area listed during the duration of the study.
7. Within 3 months of study entry topical treatment in the treatment area for actinic keratosis including, but not limited to imiquimond, 5- fluorouracil, diclofenac or liquid nitrogen.
8. Within 6 months of study entry treatments with Poly-L-lactic acid (PLLA; Sculptra Aesthetic) that may interfere with the evaluation of the treatment area.
9. Within 7 days of study entry use of self-tanners, excessive exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing) or expectations of any listed during the time of the study within the treatment area.
10. Any systemic disease that is not yet stabilized for at least six (6) Months prior to entering study.
11. A significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would interfere with the objectives of the study
12. Pregnant or nursing women or women planning a pregnancy during the study period.
13. Any unhealed skin lesions or wounds within the treatment area.
14. Existence of one (1) or more suspected basal cell carcinoma or squamous cell carcinoma within the treatment area.
15. Current participation or participation within 30 days prior to the start of this study in a drug or investigational device research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- Cosmetic Laser Dermatology, San Diego, California, United States

REFERENCES:
- [Derived] Wu DC, Guiha I, Goldman MP. A Prospective Pilot Clinical Trial to Evaluate the Efficacy and Safety of Topical Therapy with Ingenol Mebutate Gel 0.015% for Actinic Keratosis on an Expanded Area of the Chest. J Clin Aesthet Dermatol. 2017 Aug;10(8):31-36. Epub 2017 Aug 1. PMID 28979661

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Inggenol Mebutate: Inggenol Mebutate 0.015%
Period: Overall Study
Arm/Group | Active Inggenol Mebutate
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Active: Inggenol Mebutate 0.015%
Arm/Group | Active
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21
Lesion Count [Mean (Standard Deviation); unit: Lesions] | 11.3 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lesion Count From Baseline to Day 59
Description: The primary efficacy endpoint will be complete clearance of all clinically visible AKs and no development of any new AKs on day 59. Lesion clearance will be determined on day 59 (visit 7) by comparing pretreatment lesion count with current lesion count on day 59, with primary efficacy endpoint being clearance of all lesions in treatment field and no growth of new lesions.
Time Frame: Day 59
Measure: Mean (Standard Deviation); unit: Leasion Count
Arm/Group | Active
Number analyzed (Participants) | 20
Leasion Count | 2.7 (0.6)

ADVERSE EVENTS:
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 6/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=21)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) — Presence of Redness in treatment area at Day 59 visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT02446223/Prot_SAP_000.pdf